CLINICAL TRIAL: NCT03517501
Title: Scarlet-2: A Randomized, Double-Blind,Placebo-Controlled, Phase 3 Study to Assess The Safety And Efficacy of ART-123 in Subjects With Sepsis and Coagulopathy
Brief Title: The Safety And Efficacy of ART-123 in Subjects With Sepsis and Coagulopathy
Acronym: Scarlet2
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor will amend study design by incorporating reconfirmation of coagulopathy following discussion with FDA regarding findings from SCARLET1 study.
Sponsor: Asahi Kasei Pharma America Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AKPA 3-3002
Record Dates: First submitted 2018-04-23; First posted 2018-05-07 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-06

CONDITIONS: Sepsis and Coagulopathy
MeSH Terms: conditions — Sepsis; Hemostatic Disorders | interventions — ART123

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ART-123 (Active Comparator)
  Interventions: Drug: ART-123
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Comparator - Placebo

INTERVENTIONS:
Drug: ART-123 — Dose: 0.06 mg/kg/day up to a maximum dose of 6 mg/day for 6 days
  Other Names: human recombinant thrombomodulin
  Arms: ART-123
Drug: Placebo Comparator - Placebo — Dose: 0.06 mg/kg/day up to a maximum dose of 6 mg/day for 6 days
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate if ART-123 given to patients who have severe sepsis can decrease mortality.

DETAILED DESCRIPTION:
Study is to evaluate if ART-123 given to patients who have severe sepsis complicated by at least one organ dysfunction and coagulopathy can decrease mortality

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be receiving treatment in an ICU or in an acute care setting (e.g., Emergency Room, Recovery Room).
2. Subjects with either compelling evidence of infection OR clinical syndromes highly likely to be bacterial in origin, as follows (Please refer to Appendix B):

   1. Compelling objective evidence of bacterial infection and a known site of infection: Objective evidence would be met with a grossly purulent site of infections, Gram stain evidence, confirming a bacterial pathogen from normally sterile fluids (blood, urine, cerebrospinal fluid (CSF), peritoneal fluid, etc.), having either:

      * White Blood Cell (WBC) count greater > 12,000/mm3 or < 4,000/mm3 or > 10% bands within 36 hours of randomization OR
      * Temperature <36°C or fever >38°C
   2. Clinical syndromes highly likely to be bacterial in origin but not compelling

      * White Blood Cell (WBC) count greater > 12,000/mm3 or < 4,000/mm3 or > 10% bands within 36 hours of randomization AND
      * Temperature <36°C or fever >38°C
3. Current treatment with intravenous antibiotics for the acute bacterial infection (i.e. not prophylactic antibiotics)
4. Subjects with sepsis-associated organ dysfunction defined by at least one of the following:

   1. Cardiovascular Dysfunction defined as requiring both adequate fluid resuscitation and vasopressors* to maintain Mean Arterial Pressure (MAP) greater than or equal to (≥) 65 mmHg (implies fluid resuscitation alone does not raise MAP to ≥ 65 mmHg), with onset time being the time of vasopressors are initiated (end of surgery if initiated in surgery), with adequate fluid resuscitation defined as:

      • Intravenous administration of at least 20 mL/kg crystalloid or 10 mL/kg colloid infusion within 6 hours.

      OR

      •Central Venous Pressure (CVP) of greater than (>) 8 mmHg or Pulmonary Artery Wedge Pressure (PAWP) of greater than (>) 12 mmHg.
      * If dopamine is the only vasopressor used, the infusion rate must be greater than (>) 5 μg/kg/min (i.e., must be prescribed to support cardio-pulmonary perfusion). If vasopressin is used, it must be given in conjunction with another vasopressor.
   2. Respiratory Dysfunction is defined as the acute need for mechanical ventilation and PaO2/FiO2 ratio of <250 (or < 200 when lung is the site of infection) with onset time being time of intubation prior to first qualifying PaO2:FiO2 (if intubated for surgery and unable to extubate the qualifying time is the end of surgery), with mechanical ventilation defined as any type of ventilation administered via an endotracheal or nasotracheal tube.
5. Subjects with coagulopathy characterized by an INR >1.40 without other known etiology (e.g., anticoagulant therapy, chronic liver disease), and having an onset at the time of the first blood draw yielding a qualifying result (point of care device INR results must be confirmed by local laboratory).
6. Subjects with coagulopathy characterized by platelet count that meets any of the below criteria, and having an onset at the time of the first blood draw yielding a qualifying result.

   1. ≥ 20,000/mm3 and ≤ 30,000/mm3 that upon retesting after platelet transfusion is > 30,000/mm3 (qualifying at the time of the first blood draw yielding a result ≥ 20,000/mm3 and ≤ 30,000/mm3)
   2. > 30,000/mm3 to < 150,000/mm3
   3. > 30% decrease in platelet count within 24 hours
7. First and last qualifying criteria of sepsis associated organ dysfunction (as defined in Inclusion #4), platelet count and INR occurring in ≤ 24 hours

Exclusion Criteria:

Candidates for the study will be excluded if ANY of the following criteria are present:

1. Subject or Authorized Representative is unable or unwilling to provide informed consent (as applicable per local and country regulations)
2. Subject is pregnant (positive serum or urine human Chorionic Gonadotropin (hCG)) or breastfeeding or intends to get pregnant within 28 days of enrolling into the study
3. Subject is < 18 years of age
4. Body weight ≥ 175 kg
5. Subject is unwilling to allow transfusion of blood or blood products
6. Presence of an advance directive to withhold life-sustaining treatment (except Cardiopulmonary Resuscitation), or likely to have life support withdrawn within 24 hours of consent
7. Subject has had previous treatment with ART-123
8. Platelet count < 20,000/ mm3 for any reason, or for platelet count ≥ 20,000/mm3 and ≤ 30,000/mm3 that upon retesting after platelet transfusion does not increase > 30,000/mm3
9. Elevated INR, leukopenia, or thrombocytopenia that is not due to sepsis, (e.g. patients treated by chemotherapy agent). Please refer to Appendix C as an example of agents known to cause myelosuppression that should be evaluated as the cause of potential leukopenia or thrombocytopenia
10. Inability to randomize patients in ≤ 12 hours after meeting Inclusion # 7 (onset time requirements for sepsis associated organ dysfunction, INR, and platelet count)
11. ≤ 8 hours remaining from the end of a major surgery having a high risk of post-operative bleeding and randomization (e.g. extensive intraabdominal or intrathoracic dissection, debridement of a large surface area of tissue, complications arising during surgery, problems with hemostasis during surgery, surgeries of long duration, surgeries with large estimated blood loss).

    • Ensures all randomized surgical subjects with a high risk of post-operative bleeding can be dosed no earlier than 12 hours post-operatively, as described in Section 2.6.3. (minimum 8 hour delay before randomization and 4 hour maximum time to dose after randomization)
12. Stroke within 3 months prior to consent, trauma or major surgery within 3 months prior to consent that may increase the risk of bleeding
13. Known bleeding diatheses or anatomical anomaly that predisposes to hemorrhage (e.g. hemophilia, hereditary hemorrhagic telangiectasia, esophageal varices, arteriovenous malformation)
14. Gastrointestinal bleeding (e.g., melena, hematemesis) or genitourinary bleeding within 6 weeks prior to consent unless a corrective interventional procedure has been performed (i.e., therapeutic endoscopy), or there is evidence of complete resolution
15. Known thrombophilia or a history of deep-vein thrombosis or pulmonary embolism within 3 months prior to consent
16. Need for full dose anticoagulation therapy (other than IV unfractionated heparin discontinued > 12 hours prior to randomization), full dose or catheter directed thrombolysis, aspirin at a daily dose > 325 mg, long-acting antiplatelet drugs (e.g. clopidogrel, prasugrel, or ticagrelor), dual antiplatelet therapy, and doses of anticoagulants exceeding thromboprophylaxis doses within 72 hours prior to the first dose of study drug (see Appendix D for more detail)
17. Acute liver failure not due to sepsis, sepsis associated acute liver failure in any patient with a history of cirrhosis, Class C Chronic liver disease (Child-Pugh score of 10-15); (See Appendix E)
18. Acute pancreatitis where infection has not been documented by a positive blood or abdominal fluid culture or Gram stain consistent with bacterial infection. Also, in the opinion of the investigator the subject is at increased risk for developing hemorrhagic pancreatitis over the duration of the study
19. Acute renal failure not due to sepsis or chronic renal failure requiring chronic RRT (Renal Replacement Therapy)
20. Imminent death or anticipated life expectancy < 90 days for any reason other than the acute sepsis
21. Participation in another research study involving an investigational agent within 30 days prior to consent, or projected study participation before the Day 29 assessment post randomization
22. Confirmed or suspected endocarditis, malaria, Pneumocystis jiroveci pneumonia, or viral infections associated with hemorrhage (e.g. dengue fever, lassa, ebola, Bolivian) during the current admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
28 day | 28 days
  All-cause mortality

SECONDARY OUTCOMES:
3 months | 3 months
  Follow up of all-cause mortality
Resolution of organ dysfunction through 28 days as measured by: | 28 days
  Shock free and alive days
Resolution of organ dysfunction through 28 days as measured by: | 28 days
  ventilator free and alive days
Resolution of organ dysfunction through 28 days as measured by: | 28 days
  dialysis free and alive days
6 and 12 months | 6 or 12 months
  Follow-up of all-cause mortality at

CONTACTS AND LOCATIONS:
Overall Officials: David Fineberg, MD, Study Director — Asahi Kasei Pharma America

IPD SHARING:
Plan to Share IPD: No